CLINICAL TRIAL: NCT03873415
Title: Assessment of Regional Gastrointestinal Absorption of BMS-986165 Using Pharmacoscintigraphic Evaluation in Healthy Male Subjects
Brief Title: Assessment of Gut Absorption of Experimental Medication BMS-986165 in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-019
Record Dates: First submitted 2019-02-04; First posted 2019-03-13 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Formulation A (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation B (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation C (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation D (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation E (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation F (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation G (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165
- Formulation H (Experimental): Dosage formulation and area of release varies between arms
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral administration

SUMMARY:
The purpose of this study is to evaluate sites of gut absorption of BMS-986165 in males

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body mass index of 18.0 to 32.0 kg/m2, inclusive, and weight ≥ 50 kg, at screening
* Estimated glomerular filtration rate (eGFR) > 80 mL/min/1.732 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) disease of the gut that, in the opinion of the Investigator or Medical Monitor, could impact upon the absorption of study drug
* Acute diarrhea, or constipation within 3 weeks prior to randomization
* Any major surgery within 4 weeks of randomization

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986165 following Treatments A, B, C, and D | Determined over 5 days
Time of maximum observed plasma concentration (Tmax) of BMS-986165 following Treatments A, B, C, and D | Determined over 5 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986165 following Treatments A, B, C, and D | Determined over 5 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-986165 following Treatments A, B, C, and D | Determined over 5 days
Apparent plasma elimination half-life (T-HALF) of BMS-986165 following Treatments A, B, C, and D | Determined over 5 days

SECONDARY OUTCOMES:
Vital signs of body temperature | Up to 60 days
Pulse rate | Up to 60 days
Physical examination | Up to 60 days
Incidence of adverse events (AE) | Up to 90 days
Incidence of serious adverse events (SAE) | Up to 90 days
Vital sign of respiratory rate | Up to 60 days
Vital sign of supine blood pressure | Up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Scintipharma, Lexington, Kentucky, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm